CLINICAL TRIAL: NCT02370810
Title: CBT-based Internet Intervention for Adults With Tinnitus in the United Kingdom: A Randomise Controlled Trial
Brief Title: A CBT-based Internet Intervention for Adults With Tinnitus in the United Kingdom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Eldre Beukes, Mrs Eldre Wiida Beukes, Anglia Ruskin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARU-0115
Record Dates: First submitted 2015-02-03; First posted 2015-02-25 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Tinnitus
Keywords: tinnitus treatment, internet-intervention, CBT
MeSH Terms: conditions — Tinnitus; Color Vision Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): CBT-based internet-intervention for tinnitus The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8 week long e-learning intervention, with new modules introduced weekly and assignments given to practice techniques learnt.
  Interventions: Behavioral: CBT-based internet-intervention for tinnitus
- weekly check-in group with delayed treatment (Other): will complete weekly measures and commence the treatment once the experimental group completes the intervention
  Interventions: Behavioral: CBT-based internet-intervention for tinnitus

INTERVENTIONS:
Behavioral: CBT-based internet-intervention for tinnitus — The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8 week long e-learning intervention, with new modules introduced weekly and assignments given to practice techniques learnt.
  Other Names: iCBT

SUMMARY:
The purpose of this study is to determine the feasibility and effectiveness of a CBT-based internet intervention for adults with tinnitus in the United Kingdom

DETAILED DESCRIPTION:
Objectives Tinnitus is one of the most distressing disabilities and innovative ways of managing the related health care burden is required. A cognitive behavioural therapy (CTB) based internet intervention (iCBT) has been developed in Europe to improve access to tinnitus treatments. This study aims to determine the feasibility and effectiveness of iCBT in reducing the impact associated with tinnitus in the United Kingdom (UK). It furthermore, aims to establish for which subgroups of tinnitus suffers this iCBT intervention would be a suitable intervention.

Design A two-armed Randomized Control Trial (RCT), with a one year follow-up design will be used to evaluate the effectiveness iCBT on tinnitus distress Setting: This will be an internet-based study for adults with tinnitus living in the UK

Participants: Eligible participants will include adults with tinnitus for a minimum period of 3 months with internet access and no major medical or psychiatric conditions. 70 participants will be recruited for each group and will be randomly assigned using a computer generated randomization schedule by an independent research assistant after being pre-stratified for age and tinnitus severity.

Intervention: The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8 week long e-learning intervention, with new modules introduced weekly and assignments given to practice techniques learnt.

Outcome measures: The main outcome measure is the Tinnitus Functional Index. Secondary outcome measures are the Tinnitus Handicap Inventory- Screening version and self-reported measures for insomnia, hearing disability, cognitive functioning, hyperacusis, anxiety and depression and quality of life.

Hypothesis: If this intervention proves feasible it is and effective, it may have implications for the way tinnitus suffers are managed in the UK. It may be that a subset of tinnitus suffers can be managed though an e-learning treatment program, freeing up services for those with more severe problems that need face to face treatment.

ELIGIBILITY:
Inclusion Criteria

Participant's eligibility for the study is as follows:

1. Aged 18 years and over living in the UK
2. The ability to read and type in English
3. No barriers to using a computer (e.g. significant fine motor control or visual problems)
4. Internet and e-mail access, and the ability to use these
5. Commitment to completing the programme
6. Completion of the online screening and outcome questionnaires
7. Agreeing to participate in either group and be randomized to one of these groups
8. Understanding and working towards the end goal of reducing the impact and distress of tinnitus, although the strength of the tinnitus may remain the same
9. Be available for 12 months after starting the study to complete a 1 year follow-up questionnaire
10. Suffering with tinnitus for a minimum period of 3 months
11. Tinnitus outcome measure scores indicating the need for tinnitus care (26 or above on the Tinnitus Functional Index)

Exclusion Criteria

1. Reporting any major medical or psychiatric conditions
2. Reporting pulsatile, objective or unilateral tinnitus, which have not been investigated medically
3. Tinnitus as a consequence of a medical disorder, still under investigation
4. Undergoing any tinnitus therapy concurrently to partaking in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Allen, Study Chair — Anglia Ruskin University
Locations (1):
- Vision and hearing Sciences, Anglia Ruskin Univeristy, Cambridge, United Kingdom

REFERENCES:
- [Derived] Rodrigo H, Beukes EW, Andersson G, Manchaiah V. Internet-based cognitive-behavioural therapy for tinnitus: secondary analysis to examine predictors of outcomes. BMJ Open. 2021 Aug 20;11(8):e049384. doi: 10.1136/bmjopen-2021-049384. PMID 34417217
- [Derived] Beukes EW, Baguley DM, Allen PM, Manchaiah V, Andersson G. Audiologist-Guided Internet-Based Cognitive Behavior Therapy for Adults With Tinnitus in the United Kingdom: A Randomized Controlled Trial. Ear Hear. 2018 May/Jun;39(3):423-433. doi: 10.1097/AUD.0000000000000505. PMID 29095725
- [Derived] Beukes EW, Manchaiah V, Allen PM, Baguley DM, Andersson G. Internet-based cognitive behavioural therapy for adults with tinnitus in the UK: study protocol for a randomised controlled trial. BMJ Open. 2015 Sep 23;5(9):e008241. doi: 10.1136/bmjopen-2015-008241. PMID 26399571

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: CBT-based internet-intervention for tinnitus The intervention offered was a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It was an 8 week long e-learning intervention, with new modules introduced weekly and assignments given to practice techniques learnt.
- Control Group: During the active intervention phase the control group completed weekly measures and commenced the treatment once the experimental group completed the intervention (delayed treatment) paradigm
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 73 | 73
Completed | 50 | 54
Not Completed | 23 | 19

BASELINE CHARACTERISTICS:
Population: There were 3 more participants recruited per group (73 instead of 70) in case of additional drop-outs
Groups:
- Weekly check-in Group: will complete weekly measures and commence the treatment once the experimental group completes the intervention
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Weekly check-in Group | Total
Number analyzed (Participants) | 73 | 73 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.82 (12.15) | 54.31 (13.50) | 55.57 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 40 | 70
  Male | 43 | 33 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Tinnitus Severity at baseline [Mean (Standard Deviation); unit: Score on a scale (0-100)] — Measure Description: A measure of tinnitus severity. Measured on a scale of 0 to 100. Lower scores indicate less severe tinnitus. A score of 25 or higher indicates the need for an intervention. A score of 50 or above indicates severe tinnitus. If post-intervention scores are lower than baseline it indicates an improvement.
  Score on a scale (0-100) | 59.8 (18.0) | 59.2 (19.0) | 59.5 (18.4)

OUTCOME MEASURES:

1. Primary Outcome: The Tinnitus Functional Index
Description: Measure of how severe the tinnitus is Units of measurement: scores on a scale Abbreviation TFI Minimal value: 0 Maximum value 100 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat paradigm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline score | 59.79 (17.95) | 59.18 (18.96)
  8 weeks Post treatment score | 38.67 (24.26) | 53.72 (19.38)

2. Secondary Outcome: Tinnitus Handicap Inventory-screening Version
Description: Measure of tinnitus severity to use as a weekly measure Measure of how severe the tinnitus is Units of measurement: scores on a scale Abbreviation THI-S Minimal value: 0 Maximum value 40 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 22.88 (8.23) | 23.48 (8.86)
  8 weeks Post-intervention | 14.22 (10.79) | 20.68 (8.96)

3. Secondary Outcome: Insomnia Severity Index
Description: Measure of sleep problems Measure of how severe the tinnitus is Units of measurement: scores on a scale Abbreviation ISI Minimal value: 0 Maximum value 28 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline | 12.34 (6.9) | 13.52 (7.16)
  8 weeks Post-intervention | 8.6 (6.83) | 12.44 (7.21)

4. Secondary Outcome: Cognitive Failures Questionnaire
Description: Measure of how cognitive difficulties such as concentration and memory Units of measurement: scores on a scale Minimal value: 0 Maximum value 100 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  Baseline score | 38.05 (16.67) | 44.52 (18.34)
  8 weeks post intervention score | 39.97 (15.34) | 41.3 (16.73)

5. Secondary Outcome: Satisfaction With Life
Description: Quality of life measure Units of measurement: scores on a scale Minimal value: 5 Maximum value 35 Higher score is a better outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  8 weeks Post-intervention | 18.34 (6.73) | 16.17 (6.29)
  Baseline Score | 16.77 (6.31) | 16.38 (6.03)

6. Secondary Outcome: Patient Health Questionnaire
Description: Measure of signs of depressive disorders Units of measurement: scores on a scale Minimal value: 0 Maximum value 28 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  8 weeks Post-intervention | 5.89 (6.13) | 7.75 (5.22)
  Baseline | 7.88 (5.56) | 8.11 (5.92)

7. Secondary Outcome: Generalised Anxiety Disorder
Description: Measure of anxiety disorder and traits Units of measurement: scores on a scale Minimal value: 0 Maximum value 21 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: intention to treat anlaysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  Post-intervention | 5.50 (5.21) | 6.87 (4.85)
  Baseline | 7.58 (5.51) | 7.21 (5.64)

8. Secondary Outcome: Hyperacusis Questionnaire
Description: Measure of abnormal sound sensitivity Units of measurement: scores on a scale Minimal value: 0 Maximum value 42 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  Post-intervention | 16.30 (9.9) | 19.49 (9.78)
  Baseline | 19.04 (7.82) | 19.27 (9.19)

9. Secondary Outcome: Hearing Handicap Inventory- Screening Version
Description: Measure of hearing difficulties or hearing disability using a screening tool Units of measurement: scores on a scale Minimal value: 0 Maximum value 40 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Weekly check-in Group
Number analyzed (Participants) | 73 | 73
score on a scale
  8 week sPost-intervention | 15.31 (12.13) | 17.90 (10.47)
  Baseline Score | 17.26 (11.71) | 18.44 (11.06)

ADVERSE EVENTS:
Time Frame: 8 weeks post intervention and 1 year post intervention. Data collected: All-Cause Mortality: Deaths related to the study Serious Adverse Events: a severe increase in tinnitus distress; anxiety or depression related to the study Other Adverse Events: A severe increase in insomnia, hyperacusis or hearing handicap
Description: All-Cause Mortality: Deaths related to the study Serious Adverse Events: a severe increase in tinnitus distress; anxiety or depression related to the study Other Adverse Events: A severe increase in insomnia, hyperacusis or hearing handicap
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73
Other Adverse Events (participants affected / at risk) | 0/73 | 0/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=73) | Control Group (N=73)
Higher level of anxiety (General disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Participants were recruited from the general public due to interest in undertaking an Internet-intervention and not from a clinical setting. The demographical distribution showed more male participants, a slightly higher mean age distribution and longer tinnitus duration than those reported by previous iCBT trials on tinnitus. Second, the likelihood of type I errors cannot be excluded due to multiplicity of testing. Third, not all participants completed the outcome measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02370810/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02370810/ICF_001.pdf